CLINICAL TRIAL: NCT06289491
Title: Randomized Trial of Hydrus Microstent Versus Goniotomy
Brief Title: A Trial of Hydrus Microstent Versus Goniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Michael M. Lin, MD, Assistant Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000544
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Glaucoma, Open-Angle
Keywords: Incisional goniotomy; Excisional goniotomy; Hydrus Microstent; Goniotomy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Hydrus Microstent (Experimental)
  Interventions: Procedure: Hydrus Microstent
- Incisional goniotomy (Experimental)
  Interventions: Procedure: Incisional goniotomy
- Excisional goniotomy (Experimental)
  Interventions: Procedure: Excisional goniotomy

INTERVENTIONS:
Procedure: Hydrus Microstent — Patients will have a Hydrus Microstent inserted into the canal of Schlemm at the time of cataract surgery
  Arms: Hydrus Microstent
Procedure: Incisional goniotomy — Patients will have incisional goniotomy to open the trabecular meshwork with a Sinskey hook at the time of cataract surgery
  Arms: Incisional goniotomy
Procedure: Excisional goniotomy — Patients will have excisional goniotomy to remove the trabecular meshwork with a Kahook Dual Blade at the time of cataract surgery
  Arms: Excisional goniotomy

SUMMARY:
The goal of this clinical trial is to evaluate the comparative efficacy and safety of Hydrus Microstent, incisional goniotomy, and excisional goniotomy when combined with cataract surgery in patients with mild and moderate open-angle glaucoma. The main questions it aims to answer are:

* How do the intraocular pressure lowering effects of these three microinvasive glaucoma surgeries compare?
* How do the safety profiles of these three microinvasive glaucoma surgeries compare?

Participants will be randomized to one of these three microinvasive glaucoma surgeries in combination with cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract planned for surgery
* Mild to moderate open-angle glaucoma, including pigmentary glaucoma and pseudoexfoliation glaucoma
* Mild stage glaucoma includes glaucomatous optic neuropathy and visual field mean deviation better than -6.0 dB, with no points in the central 5 degrees <15 dB
* Moderate stage glaucoma includes: 1) glaucomatous optic neuropathy and visual field mean deviation equal to or worse than -6.0 dB but no worse than -12.0 dB and no central 5 degree points <15 dB or 2) mean deviation -12.0 dB or better with 1 central 5 degree point <15 dB
* Medicated IOP between 10 to 31 mm Hg, inclusive, at time of decision for surgery
* Willing and able to understand and provide informed consent
* Willing and able to attend postoperative examinations per protocol schedule

Exclusion Criteria:

* Prior argon laser trabeculoplasty, laser peripheral iridotomy, incisional glaucoma surgery, or cyclophotocoagulation
* Selective laser trabeculoplasty within 90 days of study enrollment
* Iridotrabecular contact for 180 degrees or greater
* Peripheral anterior synechiae in nasal or inferior angle
* Best corrected visual acuity worse than 20/200
* Phacodonesis on pre-operative examination
* Vitreous in anterior chamber on pre-operative examination
* Nanophthalmos
* Anti-platelet and anticoagulant medications other than aspirin 81mg daily
* Active treatment for another ophthalmic condition in either eye (e.g., anti-VEGF injections, steroids for corneal transplant)
* Abnormality in study eye that could affect tonometry
* Glaucoma diagnosis other than the above
* Normal tension glaucoma
* Conditions that can cause elevated episcleral venous pressure (e.g., Sturge-Weber syndrome, Graves disease, retrobulbar tumor)
* History of uveitis in either eye
* Inability to complete gonioscopy examination
* Use of oral steroids within 90 days or anticipated use of oral steroids
* Oral medications that can affect IOP, including oral carbonic anhydrase inhibitors such as acetazolamide and methazolamide
* History of steroid-associated IOP elevation
* Medically unfit for attending planned study visits
* Involvement in another interventional research study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 3 years
Intraocular pressure-lowering medications | 3 years

SECONDARY OUTCOMES:
Surgical complications | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No